CLINICAL TRIAL: NCT01180192
Title: Phase 3 Study of Postpartum Oxygen Inhalation for the Treatment of Postpartum Haemorrhage
Brief Title: Postpartum Oxygen Inhalation for the Treatment of Postpartum Haemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Bakirkoy Women's and Children's Teaching Hospital, Department of Obstetrics and Gynecology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: gungorduk09
Record Dates: First submitted 2010-08-09; First posted 2010-08-12 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2010-05

CONDITIONS: Postpartum Hemorrhage
Keywords: blood loss; oxygen inhalation
MeSH Terms: conditions — Postpartum Hemorrhage; Hemorrhage | interventions — Oxygen

ARMS (1):
- oxygen (Experimental)
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: oxygen — either 8 L/minute O2 via face mask for 2 hours
  Other Names: Women were randomized to receive either 8 L/minute O2 via face mask for 2 hours or breathed room air at the end of second stage of labor.

SUMMARY:
In the aetiology of postpartum uterine atony, hypoxia is considered an important factor although some suggest that peripheral oxygen saturation is not influenced by oxygen inhalation in women during the first and second stages of labor. Enhancing oxygen delivery to myometrium through additional inhaled oxygen may improve uterine contractions. Therefore, it is reasonable to consider that oxygen inhalation may promote myometrial contraction and prevent postpartum haemorrhage (PPH) due to uterine atony. The tendency for the uterus to relax in women encountering respiratory problems immediately after cesarean section under general anaesthesia further strengthened this theory.

The aim of this study was to evaluate the effectiveness of oxygen inhalation immediately after vaginal delivery on blood loss. The investigators hypothesized that inhaled oxygen helps to maintain uterine retraction during immediate postpartum period and hence reduces vaginal blood loss.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 37 and 42 weeks;
* singleton pregnancy;
* live fetus;
* cephalic presentation;
* neonatal birth weight of 2500-4500 g;
* parity between one and five;
* maternal age < 35 years old;
* vaginal birth

Exclusion Criteria:

* blood pressure ≥ 140/90mmHg;
* placenta previa;
* placental abruption;
* a history of any bleeding during pregnancy;
* a history of curettage;
* cesarean section or any uterine scar;
* a history of postpartum hemorrhage;
* polyhydramnios;
* signs or symptoms of maternal infection;
* known uterine anomalies;
* history of any drug use during labor;
* abnormal placentation;
* coagulation defects;
* instrumental deliveries;
* hemoglobin concentration < 8 g/dL;
* history of anticoagulant drugs;
* beta-mimetic medications during pregnancy;
* prolongation of the first stage of labor > 15 hours

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the amount of blood loss in the third and fourth stages of labor. | two hours
  The volume of blood loss was measured by weighing a sheet soaked from the end of the delivery to 2h after birth. Because it is important to collect the blood accurately, we used a specially designed operating sheet and an electronic scale to weigh all the material (with a 1 g deviation range). The quantity of blood (ml) = (weight of used materials - weight of materials prior to use)/1.05. Hemoglobin concentration was estimated on admission and 24 h after delivery

SECONDARY OUTCOMES:
incidences of Postpartum Haemorrhage (PPH) (≥500 ml) | two hours
  The volume of blood loss was measured by weighing a sheet soaked from the end of the delivery to 2h after birth. Because it is important to collect the blood accurately, we used a specially designed operating sheet and an electronic scale to weigh all the material (with a 1 g deviation range). The quantity of blood (ml) = (weight of used materials - weight of materials prior to use)/1.05.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Women's and Children's Teaching Hospital, Istanbul, Turkey (Türkiye)